CLINICAL TRIAL: NCT00314210
Title: A Multi-Centre,Double-Blind,Randomised-Withdrawal,Parallel-Group, Placebo-Controlled Phase III Study of the Efficacy and Safety of Quetiapine SR as Monotherapy in the Maintenance Treatment of Patients With GAD Following an Open-Label Stabilisation Period
Brief Title: Safety and Efficacy Maintenance Study of Quetiapine SR to Treat GAD Patients.
Acronym: PLATINUM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1448C00012; EUDRACT Number: 2005-005055-18
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Anxiety Disorders
Keywords: Generalised Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder

INTERVENTIONS:
Drug: Quetiapine SR

SUMMARY:
The primary objective of this study is to evaluate the efficacy of quetiapine SR compared to placebo in increasing time from randomisation to an anxiety event in patients with generalised anxiety disorder (GAD).

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be male or female, 18 to 65 years of age (inclusive), with a diagnosis of GAD according to DSM-IV criteria 300.02 as assessed by the MINI.

Exclusion Criteria:

* Patients suffering from depressive symptoms, defined as having a Montgomery-Åsberg Depression Rating Scale (MADRS) total score of 17 or more at the enrolment visit, will be excluded from participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575
Dates: Start 2006-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Time from randomisation to occurrence of an anxiety event

SECONDARY OUTCOMES:
Occurrence of an anxiety event
Change from randomisation in HAM-A/CGI-S scores
In HAM-A psychic/somatic anxiety factor scores
In MADRS total score and in MADRS item 10 score (suicidal thought)
Change in Patient Reported Outcomes (PRO): QLESQ/PSQ/SDS

CONTACTS AND LOCATIONS:
Overall Officials: Martin Brecher, MD, Study Director — AstraZeneca
Locations (114):
- United States (56):
  - Research Site, Mesa, Arizona
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Fresno, California
  - Research Site, La Mesa, California
  - Research Site, Oceanside, California
  - Research Site, Redlands, California
  - Research Site, Coral Springs, Florida
  - Research Site, DeLand, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Gainsville, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, North Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Saint Petersberg, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Libertyville, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Lafayette, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Prairie Village, Kansas
  - Research Site, Owensboro, Kentucky
  - Research Site, Paducah, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Glen Burnie, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Cambridge, Massachusetts
  - Research Site, Pittsfield, Massachusetts
  - Research Site, Saint Charles, Missouri
  - Research Site, Piscataway, New Jersey
  - Research Site, Cedarhurst, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, Avon Lake, Ohio
  - Research Site, Beechwood, Ohio
  - Research Site, Cincinnati, Ohio
  - Research SIte, Middleburg Heights, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Allentown, Pennsylvania
  - Research Site, Havertown, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, North Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, DeSoto, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Midvale, Utah
  - Research Site, Richmond, Virginia
- Australia (5):
  - Research Site, Brisbane, Queensland
  - Research Site, Everton Park, Queensland
  - Research Site, West Burleigh, Queensland
  - Research Site, Malvern, Victoria
  - Research Site, Prahran, Victoria
- Canada (9):
  - Research Site, Edmonton, Alberta
  - Research Site, Bathurst, New Brunswick
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Orléans, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Montreal, Quebec
- Finland (7):
  - Research Site, Helsinki
  - Research Site, Joensuu
  - Research Site, Kuopio
  - Research Site, Oulu
  - Research Site, Pori
  - Research Site, Seinäjoki
  - Research Site, Turku
- Germany (9):
  - Research Site, Berlin
  - Research Site, Göttingen
  - Research Site, Jena
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Naumburg
  - Research Site, Nuremberg
  - Research Site, Schwerin
  - Research Site, Siegen
- Hungary (6):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Kecskemét
  - Research Site, Nyíregyháza
- Indonesia (2):
  - Research Site, Bandung, West Java
  - Research Site, Jakarta
- Philippines (5):
  - Research Site, Cebu City
  - Research Site, Davao City
  - Research Site, Mandaluyong
  - Research Site, Manila
  - Research Site, Quezon City
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Saratov
- Research Site, Seoul, South Korea
- United Kingdom (11):
  - Research Site, Reading, Berkshire
  - Research Site, Crawley, West Sussex
  - Research Site, Blackpool
  - Research Site, Bolton
  - Research Site, Cardiff
  - Research Site, Chorley
  - Research Site, Coventry
  - Research Site, Glasgow
  - Research Site, Hamilton
  - Research Site, Liverpool
  - Research Site, Manchester

REFERENCES:
- [Derived] Sheehan DV, Svedsater H, Locklear JC, Eriksson H. Effects of extended-release quetiapine fumarate on long-term functioning and sleep quality in patients with Generalized Anxiety Disorder (GAD): data from a randomized-withdrawal, placebo-controlled maintenance study. J Affect Disord. 2013 Dec;151(3):906-13. doi: 10.1016/j.jad.2013.07.037. Epub 2013 Aug 16. PMID 24135509